CLINICAL TRIAL: NCT03688672
Title: Evaluation of the Feasibility of Fitting of Apioc Contact Lenses in Adults
Brief Title: Apioc Contact Lens Feasibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lentechs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: LEN001
Record Dates: First submitted 2018-09-25; First posted 2018-09-28 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Ametropia; Myopia; Hyperopia; Astigmatism; Presbyopia
Keywords: contact lens; soft contact lens; feasibility
MeSH Terms: conditions — Refractive Errors; Myopia; Hyperopia; Astigmatism; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Apioc Lens (Other): All subjects will wear the same, Apioc Contact Lens design.
  Interventions: Device: Apioc Contact Lens Design

INTERVENTIONS:
Device: Apioc Contact Lens Design — Novel soft contact lens design.

SUMMARY:
This clinical trial will document the feasibility of the Apioc lens design by assessing which lens shape parameters yield successful on-eye-fit and movement of the Apioc contact lens design and evaluate the subjectively-reported comfort of the Apioc contact lens design.

DETAILED DESCRIPTION:
This is a one-site, non-dispensing clinical trial using the Apioc contact lens design. This soft contact lens study will determine the feasibility of this design by determining which parameters of the shape of the Apioc Contact Lens design will yield a successful fit across subjects. We will also determine the percentage of subjects who can be successfully fitted with the Apioc Contact Lens Design. Because the feasibility of the lens design may be dependent upon age, a total of 50 subjects (10 subjects each across 5 decades of life) will complete the study. The data will be collected in a single visit for most subjects. A few subjects may be asked to return for a second visit if additional contact lens parameters need to be ordered to achieve a successful fit. The key assessments for this study will be demonstration of feasibility of fit, documentation of movement in all gazes, including translation, and subjective reports of comfort. Subjects will only wear contact lenses while in the office.

ELIGIBILITY:
Inclusion Criteria:

1. Thirty subjects will be at least 40 years of age and no more than 60 years of age. Ten subjects will be at least 18 years of age and no more than 29 years of age. Ten subjects will be at least 30 years of age and no more than 39 years of age.
2. The subject must have ≤ 1.50 D of corneal astigmatism.
3. The subject should have clear, healthy corneas.
4. The subject should have a normal, healthy conjunctiva in both eyes.
5. The subject should be free of active ocular disease. Refractive error and presbyopia are permitted.
6. The subject must provide written informed consent.
7. The subject must appear willing and able to adhere to the instructions set forth in this protocol.

Exclusion Criteria:

1. No irregular corneal astigmatism is permitted.
2. No pterygia or corneal scarring that would interfere with contact lens wear.
3. No pinguecula or other conjunctival thickness abnormalities are permitted that would interfere with contact lens wear.
4. The subject should not be using any ocular pharmaceutical treatments, including artificial tears in the two weeks prior to the examination.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Vertical Movement of Contact Lens in Downgaze | After 15 minutes of on-eye settling
  Vertical movement of the contact lens relative to the eye in downgaze in millimeters.

SECONDARY OUTCOMES:
Movement of contact lens with blink | After 15 minutes of on-eye settling
  Movement of contact lens in straight-ahead gaze with a blink in millimeters.
Visual Acuity | After 15 minutes of on-eye settling
  logMAR visual acuity at 40 cm through the contact lens with distance correction in trial frame over the Apioc contact lens.
Comfort questionnaire | After 15 minutes of on-eye settling
  Subjects will be asked to assess the comfort of each lens by marking an "X" on a line between 0 and 100.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Wagner, OD, MS, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No